CLINICAL TRIAL: NCT00306384
Title: A Long-Term, Open-Label Extension Study to Investigate the Long-Term Safety of SYR110322 (SYR-322) in Subjects With Type 2 Diabetes
Brief Title: Long-term Safety of Alogliptin in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYR-322-OLE-012; 2005-004672-20 (EudraCT Number); U1111-1113-8455 (Registry Identifier: WHO)
Record Dates: First submitted 2006-03-21; First posted 2006-03-23 (Estimated); Results first posted 2013-03-22 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-02

CONDITIONS: Diabetes Mellitus
Keywords: Glucose Metabolism Disorder; Dysmetabolic Syndrome; Type II Diabetes; Diabetes Mellitus,; Lipoatrophic; Dyslipidemia; Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus; Glucose Metabolism Disorders; Diabetes Mellitus, Type 2; Dyslipidemias | interventions — alogliptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alogliptin 12.5 mg (Experimental): Alogliptin 12.5 tablet, orally, once daily for up to 4 years.
  Interventions: Drug: Alogliptin
- Alogliptin 25 mg (Experimental): Alogliptin 25 mg tablet, orally, once daily for up to 4 years.
  Interventions: Drug: Alogliptin

INTERVENTIONS:
Drug: Alogliptin — Alogliptin tablets.
  Other Names: SYR110322; SYR-322

SUMMARY:
The purpose of this study is to evaluate the long-term safety of alogliptin, once daily (QD), following participation in 1 of 7 controlled studies in patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
SYR-322 (alogliptin) is an inhibitor of the dipeptidyl peptidase IV enzyme. Dipeptidyl peptidase IV is thought to be primarily responsible for the degradation of 2 peptide hormones released in response to nutrient ingestion, namely glucagon-like peptide-1 and glucose-dependent insulinotropic peptide. It is expected that inhibition of dipeptidyl peptidase IV will improve glycemic (glucose) control in patients with type 2 diabetes mellitus by prolonging the beneficial effects of glucagon-like peptide-1.

The rising incidence of type 2 diabetes mellitus and the limitations of the currently available treatments suggest the need for new therapies for glycemic control. Studies have been undertaken in humans that evaluated the effects of directly augmenting glucagon-like peptide-1 and glucose-dependent insulinotropic peptide levels and of inhibiting the activity of dipeptidyl peptidase IV.

This study is an extension of 7 controlled phase 3 studies of alogliptin. These phase 3 studies included 1 monotherapy study of alogliptin (SYR-322-PLC-010; NCT00286455); 4 placebo-controlled add-on studies of alogliptin, namely in combination with a sulfonylurea (SYR-322-SULF-007; NCT00286468), metformin (SYR-322-MET-008; NCT00286442), a thiazolidinedione (pioglitazone; SYR-322-TZD-009; NCT00286494), and insulin (SYR-322-INS-011; NCT00286429); 1 coadministration study with pioglitazone in combination with metformin (01-05-TL-322OPI-001; NCT00328627), and 1 coadministration study with pioglitazone (01-06-TL-322OPI-002; NCT00395512).

The end of treatment or early withdrawal visit from the preceding study will be the screening visit for this study, after which enrolled patients will be required to commit to approximately 22 additional visits at the study center.

ELIGIBILITY:
Inclusion Criteria:

* Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.
* Type 2 diabetes mellitus and was enrolled in one of the following 7 controlled Phase III studies. The study will be open to all patients who completed one of these studies through the end-of-treatment visit:

  * SYR-322-PLC-010 - NCT00286455
  * SYR-322-SULF-007 - NCT00286468
  * SYR-322-MET-008 - NCT00286442
  * SYR-322-TZD-009 - NCT00286494
  * SYR-322-INS-011 - NCT00286429
  * 01-05-TL-322OPI-001 - NCT00328627
  * 01-06-TL-322OPI-002 - NCT00395512
* Alanine aminotransferase less than or equal to 3 times the upper limit of normal and serum creatinine less than or equal to 2.0 mg per dL.
* Able and willing to monitor own blood glucose concentrations with a home glucose monitor.
* No major illness or debility that in the investigator's opinion prohibits the patient from completing the study.

Exclusion Criteria

* The occurrence of any adverse event or condition during the controlled Phase III studies, which, in the opinion of the investigator, should exclude the patient from participating in the open-label extension.
* Is required to take or intends to continue taking any disallowed medication, any prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of the study medication, including:

  * Weight-loss drugs
  * Investigational antidiabetics, additional dipeptidyl peptidase-4 (DPP-4) and glucagon-like peptide-1 (GLP 1) inhibitors
  * Incretin Mimetics,
  * Oral or systemically injected glucocorticoids.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3323 (Actual)
Dates: Start 2006-03; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: VP Biological Sciences, Study Director — Takeda
Locations (114):
- United States (62):
  - Birmingham, Alabama
  - Peoria, Arizona
  - Phoenix, Arizona
  - Anaheim, California
  - Artesia, California
  - Fresno, California
  - Los Angeles, California
  - Mission Viejo, California
  - Northridge, California
  - Orange, California
  - San Diego, California
  - Tustin, California
  - Walnut Creek, California
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Norwalk, Connecticut
  - Washington D.C., District of Columbia
  - Clearwater, Florida
  - Hollywood, Florida
  - Kissimmee, Florida
  - Longwood, Florida
  - New Port Richie, Florida
  - Ocala, Florida
  - Ocoee, Florida
  - Saint Cloud, Florida
  - Lawrenceville, Georgia
  - Honolulu, Hawaii
  - Idaho Falls, Idaho
  - Chicago, Illinois
  - Avon, Indiana
  - Elkhart, Indiana
  - Evansville, Indiana
  - Lafayette, Indiana
  - Erlanger, Kentucky
  - Baltimore, Maryland
  - Sudbury, Massachusetts
  - Chesterfield, Missouri
  - St Louis, Missouri
  - Omaha, Nebraska
  - Berlin, New Jersey
  - Burlington, North Carolina
  - Charlotte, North Carolina
  - Morehead City, North Carolina
  - Pinehurst, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnatti, Ohio
  - Dayton, Ohio
  - Tulsa, Oklahoma
  - Medford, Oregon
  - Lansdale, Pennsylvania
  - West Grove, Pennsylvania
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Simpsonville, South Carolina
  - Bristol, Tennessee
  - Cookeville, Tennessee
  - Milan, Tennessee
  - Dallas, Texas
  - San Antonio, Texas
  - Temple, Texas
  - Texarkana, Texas
  - Burlington, Vermont
- Argentina (7):
  - Buenos Aires, La Plata
  - Buenos Aires, Moron
  - Rosario, Sante Fe
  - Buenos Aires
  - Ciudadd Autonoma de Buenos Aires
  - Córdoba
  - Mar del Plata
- Brazil (6):
  - Fortaleza, Ceará
  - Curitiba, Paraná
  - Porto Alegre, Rio Grande do Sul
  - Mogi das Cruzes, São Paulo
  - Santos, São Paulo
  - São Paulo
- Santiago, Chile
- Czechia (4):
  - Ostrava
  - Prague
  - Sternberk
  - Zlín
- Santo Domingo Oeste, Dominican Republic
- Germany (10):
  - Aschaffenburg
  - Berlin
  - Frankfurt
  - Hamburg
  - Hanover
  - Munich
  - Nuremberg
  - Schwerin
  - Wiesbaden
  - Witten
- Guatemala City, Guatemala
- Netherlands (6):
  - Almere Stad
  - De Bilt
  - Geleen
  - Oud-Beijerland
  - Rotterdam
  - Zwijndrecht
- Peru (4):
  - Bellavista, Lima region
  - San Isidro, Lima region
  - Ica
  - Lima
- Poland (6):
  - Bytom
  - Kamieniec Ząbkowicki
  - Krakow
  - Lodz
  - Radom
  - Łęczyca
- South Africa (6):
  - Pretoria, Gauteng
  - Cape Town, Western Cape
  - Somerset West, Western Cape
  - Durban
  - Johannesburg
  - Parow

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients who completed 1 of the following 7 studies took part in the study at 423 investigative sites worldwide: SYR-322-PLC-010 (NCT00286455); SYR-322-SULF-007 (NCT00286468); SYR-322-MET-008 (NCT00286442); SYR-322-TZD-009 (NCT00286494); SYR-322-INS-011 (NCT00286429); 01-05-TL-322OPI-001 (NCT00328627); 01-06-TL-322OPI-002 (NCT00395512).
Pre-assignment Details: Patients who had previously completed 1 of 7 double-blind alogliptin studies were randomized (1:1) to either 12.5 or 25 mg once daily alogliptin. Patients who were rescued during their previous double-blind study in response to protocol-defined hyperglycemic rescue criteria were assigned to alogliptin 25 mg.
Groups:
- Alogliptin 12.5 mg: Participants who completed the previous double-blind study received alogliptin 12.5 tablet, orally, once daily for up to 4 years.
- Alogliptin 25 mg: Participants who completed the previous double-blind study received alogliptin 25 mg tablets orally, once daily for up to 4 years.
- Rescued: Alogliptin 25 mg: Participants rescued from the previous double-blind study received alogliptin 25 mg tablets, orally once daily for up to 4 years.
Period: Overall Study
Arm/Group | Alogliptin 12.5 mg | Alogliptin 25 mg | Rescued: Alogliptin 25 mg
Started | 1396 | 1399 | 528
Safety Set | 1395 (Patients who received at least one dose of study drug) | 1398 (Patients who received at least one dose of study drug) | 527 (Patients who received at least one dose of study drug)
Completed | 854 | 891 | 251
Not Completed | 542 | 508 | 277
Not completed — Adverse Event | 103 | 87 | 40
Not completed — Major protocol deviation | 43 | 51 | 18
Not completed — Lost to Follow-up | 57 | 41 | 35
Not completed — Voluntary withdrawal | 199 | 187 | 91
Not completed — Study termination | 1 | 0 | 1
Not completed — Pregnancy | 3 | 1 | 1
Not completed — Lack of Efficacy | 26 | 40 | 38
Not completed — Investigator discretion | 28 | 31 | 21
Not completed — Other | 80 | 70 | 32
Not completed — Site closure | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alogliptin 12.5 mg | Alogliptin 25 mg | Rescued: Alogliptin 25 mg | Total
Number analyzed (Participants) | 1396 | 1399 | 528 | 3323
Age Continuous [Mean (Standard Deviation); unit: years] | 55.8 (9.92) | 55.1 (10.21) | 53.0 (10.06) | 55.0 (10.11)
Age, Customized [Number; unit: participants]
  <65 years | 1134 | 1134 | 461 | 2729
  ≥65 years | 262 | 265 | 67 | 594
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 699 | 730 | 289 | 1718
  Male | 697 | 669 | 239 | 1605
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 8 | 3 | 2 | 13
  Asian | 120 | 108 | 32 | 260
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 1 | 3
  Black or African American | 65 | 88 | 34 | 187
  White | 1025 | 1007 | 390 | 2422
  Other | 176 | 193 | 69 | 438
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 31.42 (5.370) | 31.71 (5.266) | 32.20 (5.704) | 31.66 (5.386)
Diabetes duration [Mean (Standard Deviation); unit: years] | 6.56 (5.446) | 6.92 (5.824) | 8.35 (6.325) | 6.99 (5.784)
Previous double-blind study treatment [Number; unit: participants] — Patients from coadministration Studies 01-05-TL-322OPI-001 and 01-06-TL-322OPI-002 are presented separately; due to the complexity of treatment assignments, they were not included in the subgroups of patients previously randomized to placebo, alogliptin 12.5 mg, or alogliptin 25 mg.
  participants
    Placebo | 118 | 110 | 135 | 363
    Alogliptin 12.5 mg | 274 | 262 | 105 | 641
    Alogliptin 25 mg | 243 | 262 | 99 | 604
    Study 01-05-TL-322OPI-001 | 546 | 548 | 146 | 1240
    Study 01-06-TL-322OPI-002 | 215 | 217 | 43 | 475

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: Safety was assessed by physical examinations, clinical laboratory parameters, electrocardiogram (ECG) readings, vital sign measurements, oral temperature, and hypoglycemic events. Changes in laboratory values or ECG parameters were considered to be adverse events if they were judged to be clinically significant. A TEAE was any event that started on or after the first dose of open-label study drug and within 14 days after the last dose.
Time Frame: 4 years
Population: Safety set
Measure: Number; unit: percentage of participants
Arm/Group | Alogliptin 12.5 mg | Alogliptin 25 mg | Rescued: Alogliptin 25 mg
Number analyzed (Participants) | 1394 | 1399 | 527
percentage of participants
  Any treatment emergent adverse event (TEAE) | 87.2 | 87.1 | 84.6
  Study drug-related TEAE | 25.6 | 22.7 | 24.9
  TEAE leading to discontinuation | 7.0 | 6.1 | 7.6
  Treatment emergent serious AE | 16.7 | 16.3 | 15.7
  Study drug-related serious AE | 2.6 | 2.1 | 1.9
  Treatment-emergent deaths | 1.4 | 1.0 | 0.9

2. Secondary Outcome: Change From Baseline Over Time in Glycosylated Hemoglobin
Description: The change from Baseline in glycosylated hemoglobin (HbA1c; the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) during the study. Endpoint was defined as the last postbaseline observation collected within 7 days after the last dose of open-label study drug.
Time Frame: Baseline and Month 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42 and 45.
Population: Safety set where data were available.
Measure: Mean (Standard Deviation); unit: percent glycosylated hemoglobin
Arm/Group | Alogliptin 12.5 mg | Alogliptin 25 mg | Rescued: Alogliptin 25 mg
Number analyzed (Participants) | 1395 | 1398 | 527
percent glycosylated hemoglobin
  Baseline (n=1362, 1359, 501) | 7.21 (0.815) | 7.22 (0.814) | 9.30 (0.900)
  Week 12 change from Baseline (n=1290, 1286, 463) | 0.18 (0.635) | 0.14 (0.632) | -0.52 (1.064)
  Month 6 change from Baseline (n= 1236, 1252, 433) | 0.31 (0.859) | 0.26 (0.848) | -0.73 (1.285)
  Month 9 change from Baseline (n=1217, 1231, 413) | 0.34 (0.969) | 0.33 (0.894) | -0.78 (1.282)
  Month 12 change from Baseline (1175, 1182, 388) | 0.41 (1.010) | 0.41 (0.952) | -0.78 (1.309)
  Month 15 change from Baseline (n=1119, 1133, 374) | 0.47 (0.990) | 0.48 (1.068) | -0.75 (1.332)
  Month 18 change from Baseline (n=1111, 1095, 350) | 0.50 (1.082) | 0.50 (1.047) | -0.70 (1.320)
  Month 21 change from Baseline (n=1061, 1071, 338) | 0.52 (1.096) | 0.51 (1.070) | -0.75 (1.389)
  Month 24 change from Baseline (n=1027, 1039, 320) | 0.53 (1.111) | 0.58 (1.107) | -0.69 (1.417)
  Month 27 change from Baseline (n=991, 1002, 300) | 0.58 (1.124) | 0.58 (1.159) | -0.71 (1.349)
  Month 30 change from Baseline (n=944, 955, 281) | 0.57 (1.127) | 0.57 (1.167) | -0.78 (1.361)
  Month 33 change from Baseline (n=923, 941, 276) | 0.55 (1.181) | 0.57 (1.196) | -0.73 (1.418)
  Month 36 change from Baseline (n=882, 931, 274) | 0.54 (1.215) | 0.55 (1.141) | -0.80 (1.411)
  Month 39 change from Baseline (n=886, 913, 259) | 0.56 (1.223) | 0.56 (1.216) | -0.73 (1.431)
  Month 42 change from Baseline (n=854, 891, 252) | 0.59 (1.225) | 0.54 (1.221) | -0.78 (1.492)
  Month 45 change from Baseline (n=866, 902, 253) | 0.61 (1.250) | 0.56 (1.242) | -0.70 (1.398)
  Endpoint change from Baseline (n=1362, 1359, 501) | 1.63 (1.310) | 0.61 (1.261) | -0.42 (1.448)

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose
Description: The change from Baseline in fasting plasma glucose (FPG) at the last post-baseline observation, collected within 7 days after the last dose of open-label study drug.
Time Frame: Baseline and Year 4
Population: Safety set where data were available.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg | Alogliptin 25 mg | Rescued: Alogliptin 25 mg
Number analyzed (Participants) | 1388 | 1386 | 517
mg/dL
  Baseline | 144.4 (41.64) | 142.6 (39.41) | 215.3 (60.25)
  Change from Baseline | 14.8 (56.25) | 14.9 (53.46) | -26.4 (84.51)

4. Secondary Outcome: Percentage of Participants With Marked Hyperglycemia
Description: Marked Hyperglycemia is defined as fasting plasma glucose greater than or equal to 200 mg/dL (≥11.10 mmol/L).
  The Month 42 to Month 45 interval includes all marked hyperglycemic episodes occurring on or after Day 1247 (a 203-day visit window).
Time Frame: Randomization up to 4 years.
Population: Safety set where data were available.
Measure: Number; unit: percentage of participants
Arm/Group | Alogliptin 12.5 mg | Alogliptin 25 mg | Rescued: Alogliptin 25 mg
Number analyzed (Participants) | 1395 | 1398 | 527
percentage of participants
  Day 1 to <Week 2 (n=1299, 1290, 481) | 9.1 | 8.0 | 55.5
  Week 2 to <Week 4 (n=1286, 1306, 481) | 11.5 | 10.2 | 45.9
  Week 4 to <Week 8 (n=1303, 1331, 490) | 9.2 | 11.0 | 46.1
  Week 8 to <Week 12 (n=1331, 1347, 495) | 11.5 | 10.8 | 41.0
  Week 12 to <Month 6 (n=1329, 1338, 480) | 12.0 | 11.6 | 39.4
  Month 6 to <Month 9 (n=1286, 1289, 448) | 12.8 | 10.7 | 36.8
  Month 9 to <Month 12 (n=1252, 1260, 425) | 11.4 | 12.9 | 32.5
  Month 12 to <Month 15 (n=1210, 1217, 409) | 13.1 | 13.0 | 29.3
  Month 15 to <Month 18 (n=1157, 1166, 389) | 12.7 | 13.8 | 27.8
  Month 18 to <Month 21 (n=1128, 1128, 365) | 11.7 | 11.6 | 26.8
  Month 21 to <Month 24 (n=1094,1099, 357) | 11.2 | 11.5 | 26.3
  Month 24 to <Month 27 (n=1046, 1066, 334) | 11.6 | 12.3 | 24.9
  Month 27 to <Month 30 (n=1010, 1028, 316) | 12.6 | 11.8 | 24.7
  Month 30 to <Month 33 (n=981, 988, 299) | 11.6 | 11.7 | 19.7
  Month 33 to <Month 36 (n=945, 959, 289) | 11.5 | 12.3 | 23.5
  Month 36 to <Month 39 (n=920, 949, 281) | 13.2 | 12.5 | 21.0
  Month 39 to <Month 42 (n=899, 934, 267) | 13.7 | 13.1 | 19.5
  Month 42 to Month 45 (n=889, 921, 261) | 25.5 | 23.9 | 39.1
  Overall (n= 1389, 1392, 518) | 49.7 | 50.7 | 87.6

5. Secondary Outcome: Change From Baseline in Proinsulin Level
Description: Proinsulin is a precursor to insulin, and was measured as an indicator of pancreatic function. The change from Baseline in fasting proinsulin to the last post-baseline observation, collected within 7 days after the last dose of open-label study drug.
  Note: A transcription error occurred in the reporting of 1 proinsulin value for a patient in the alogliptin 25 mg completed group, for whom a partial patient ID number was mistakenly entered as an end-of-treatment proinsulin level.
Time Frame: Baseline and Year 4
Population: Safety set where data were available.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Alogliptin 12.5 mg | Alogliptin 25 mg | Rescued: Alogliptin 25 mg
Number analyzed (Participants) | 1277 | 1263 | 393
pmol/L
  Baseline | 26.1 (25.99) | 25.4 (30.28) | 40.2 (36.47)
  Change from Baseline | 4.1 (27.09) | 39.7 (1243.37) | -3.3 (31.45)

6. Secondary Outcome: Change From Baseline in Insulin Level
Description: The change from Baseline in fasting insulin at the last post-baseline observation, collected within 7 days after the last dose of open-label study drug.
Time Frame: Baseline and Year 4
Population: Safety set where data was available. Does not include patients enrolled in Protocol 01-05-TL-OPI322-001 or Protocol 01-06-TL-OPI322-002.
Measure: Mean (Standard Deviation); unit: μIU/mL
Arm/Group | Alogliptin 12.5 mg | Alogliptin 25 mg | Rescued: Alogliptin 25 mg
Number analyzed (Participants) | 537 | 526 | 212
μIU/mL
  Baseline | 15.19 (9.898) | 15.50 (12.608) | 18.64 (15.845)
  Change from Baseline | 2.45 (42.706) | 2.13 (16.496) | 5.62 (23.197)

7. Secondary Outcome: Change From Baseline in C-peptide Level
Description: C-peptide is a byproduct created when the hormone insulin is produced and is measured by a blood test. Change from Baseline to the last post-baseline observation, collected within 7 days after the last dose of open-label study drug.
Time Frame: Baseline and Year 4
Population: Safety set where data was available. Patients enrolled in Protocol 01-05-TL-OPI322-001 or Protocol 01-06-TL-OPI322-002 are not included.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Alogliptin 12.5 mg | Alogliptin 25 mg | Rescued: Alogliptin 25 mg
Number analyzed (Participants) | 615 | 615 | 322
ng/mL
  Baseline | 3.406 (1.5115) | 3.323 (1.5945) | 3.572 (1.7531)
  Change from Baseline | -0.471 (1.6464) | -0.439 (1.2783) | -0.641 (1.5804)

8. Secondary Outcome: Change From Baseline in Body Weight
Description: Change from Baseline in body weight to the last post-baseline observation collected within 7 days after the last dose of open-label study drug.
Time Frame: Baseline and Year 4
Population: Safety set for whom data was available.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Alogliptin 12.5 mg | Alogliptin 25 mg | Rescued: Alogliptin 25 mg
Number analyzed (Participants) | 1387 | 1385 | 518
kg
  Baseline | 86.12 (19.376) | 86.61 (19.185) | 88.62 (20.947)
  Change from Baseline | -0.64 (5.283) | -0.61 (5.428) | 0.25 (5.036)

9. Secondary Outcome: Percentage of Participants With a Clinical Response
Description: Clinical response was defined based on the absolute value of HbA1c meeting one of two clinical targets at any post-baseline visit:
  * HbA1c ≤6.5%;
  * HbA1c ≤7.0%.
Time Frame: Weeks 2, 4, 8, 12, every 3 months up to 4 years, and 1 Day after final dose.
Population: Safety set.
Measure: Number; unit: percentage of participants
Arm/Group | Alogliptin 12.5 mg | Alogliptin 25 mg | Rescued: Alogliptin 25 mg
Number analyzed (Participants) | 1395 | 1398 | 527
percentage of participants
  HbA1c ≤6.5% | 34.8 | 34.1 | 11.0
  HbA1c ≤7.0% | 64.1 | 65.5 | 27.1

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (AEs) were defined as any AEs that started on or after the date of the first dose of open-label study drug and within 14 days after the date of the last dose of open-label study drug.
Description: At each study visit, the investigator assessed whether any events had occurred. Participants could report events at any other time during the study.
Arm/Group | Alogliptin 12.5 mg | Alogliptin 25 mg | Rescued: Alogliptin 25 mg
Serious Adverse Events (participants affected / at risk) | 233/1394 | 228/1399 | 83/527
Other Adverse Events (participants affected / at risk) | 876/1394 | 898/1399 | 333/527
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alogliptin 12.5 mg (N=1394) | Alogliptin 25 mg (N=1399) | Rescued: Alogliptin 25 mg (N=527)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 7 | 11 | 4
Coronary artery disease (Cardiac disorders) | 5 | 7 | 5
Myocardial infarction (Cardiac disorders) | 5 | 6 | 4
Angina pectoris (Cardiac disorders) | 5 | 5 | 2
Angina unstable (Cardiac disorders) | 6 | 3 | 2
Myocardial ischaemia (Cardiac disorders) | 7 | 3 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 4 | 1
Acute coronary syndrome (Cardiac disorders) | 2 | 1 | 2
Cardiac failure congestive (Cardiac disorders) | 0 | 2 | 2
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 2 | 1
Cardiac failure (Cardiac disorders) | 1 | 2 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 2 | 0
Atrioventricular block complete (Cardiac disorders) | 2 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 2 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 1 | 1
Pericardial effusion (Cardiac disorders) | 2 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 1
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 0 | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0 | 0
Congestive cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Coronary artery insufficiency (Cardiac disorders) | 1 | 0 | 0
Hypertensive heart disease (Cardiac disorders) | 0 | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 0 | 1 | 0
MELAS syndrome (Congenital, familial and genetic disorders) | 1 | 0 | 0
Goitre (Endocrine disorders) | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 2 | 1 | 0
Retinal vein thrombosis (Eye disorders) | 0 | 2 | 0
Diabetic retinopathy (Eye disorders) | 1 | 0 | 0
Glaucoma (Eye disorders) | 0 | 0 | 1
Iridocyclitis (Eye disorders) | 1 | 0 | 0
Retinal artery occlusion (Eye disorders) | 0 | 1 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 1
Vitreous haemorrhage (Eye disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 4 | 1
Inguinal hernia (Gastrointestinal disorders) | 3 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 2 | 0
Pancreatitis acute (Gastrointestinal disorders) | 3 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal hypomotility (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Hernial eventration (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis relapsing (Gastrointestinal disorders) | 0 | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Peritonitis (Gastrointestinal disorders) | 1 | 0 | 0
Rectal polyp (Gastrointestinal disorders) | 1 | 0 | 0
Rectal prolapse (Gastrointestinal disorders) | 0 | 1 | 0
Salivary duct inflammation (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 4 | 4 | 2
Chest pain (General disorders) | 1 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 2
Death (General disorders) | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 3 | 4 | 2
Cholecystitis acute (Hepatobiliary disorders) | 4 | 2 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 2 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 0
Perforation bile duct (Hepatobiliary disorders) | 0 | 1 | 0
Allergic oedema (Immune system disorders) | 1 | 0 | 0
Allergy to arthropod sting (Immune system disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 13 | 6 | 0
Cellulitis (Infections and infestations) | 4 | 3 | 4
Urinary tract infection (Infections and infestations) | 5 | 4 | 0
Erysipelas (Infections and infestations) | 2 | 3 | 0
Osteomyelitis (Infections and infestations) | 3 | 1 | 1
Diverticulitis (Infections and infestations) | 2 | 2 | 0
Gastroenteritis (Infections and infestations) | 1 | 2 | 1
Gangrene (Infections and infestations) | 2 | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 1 | 1
Abscess limb (Infections and infestations) | 1 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 2 | 0
Bronchopneumonia (Infections and infestations) | 0 | 2 | 0
Dengue fever (Infections and infestations) | 2 | 0 | 0
Diabetic foot infection (Infections and infestations) | 1 | 0 | 1
Infected skin ulcer (Infections and infestations) | 1 | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 0 | 2
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Post procedural infection (Infections and infestations) | 0 | 1 | 1
Pyelonephritis (Infections and infestations) | 0 | 2 | 0
Staphylococcal infection (Infections and infestations) | 2 | 0 | 0
Viral infection (Infections and infestations) | 1 | 0 | 1
Acquired immunodeficiency syndrome (Infections and infestations) | 0 | 1 | 0
Appendicitis perforated (Infections and infestations) | 0 | 1 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0 | 0
Cholecystitis infective (Infections and infestations) | 1 | 0 | 0
Coccidioidomycosis (Infections and infestations) | 0 | 0 | 1
Endophthalmitis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0
Giardiasis (Infections and infestations) | 0 | 1 | 0
Helicobacter gastritis (Infections and infestations) | 0 | 1 | 0
Hepatitis A (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Labyrinthitis (Infections and infestations) | 0 | 1 | 0
Lymphangitis (Infections and infestations) | 1 | 0 | 0
Nosocomial infection (Infections and infestations) | 0 | 1 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 1 | 0
Pneumococcal sepsis (Infections and infestations) | 1 | 0 | 0
Pneumonia cryptococcal (Infections and infestations) | 1 | 0 | 0
Pneumonia pneumococcal (Infections and infestations) | 1 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0
Pyelonephritis chronic (Infections and infestations) | 0 | 1 | 0
Pyoderma (Infections and infestations) | 0 | 0 | 1
Rectal abscess (Infections and infestations) | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0
Sialoadenitis (Infections and infestations) | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 0
Typhoid fever (Infections and infestations) | 0 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 1 | 0
Wound sepsis (Infections and infestations) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 1 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 3 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 3 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 2 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Tendon injury (Injury, poisoning and procedural complications) | 1 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 0 | 0
Chest injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Device occlusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Foreign body trauma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Incisional hernia, obstructive (Injury, poisoning and procedural complications) | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 3 | 3
Diabetic foot (Metabolism and nutrition disorders) | 1 | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Obesity (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypoglycaemic seizure (Metabolism and nutrition disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 6 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 6 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 | 3 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Chondromalacia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tendon calcification (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 2
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Benign neoplasm of adrenal gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Brain neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Breast cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Carcinoid tumour of the appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Central nervous system neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cervix neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Choroid melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Colon cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Focal nodular hyperplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Langerhans' cell granulomatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Oligodendroglioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Prostatic adenom (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 6 | 1 | 4
Ischaemic stroke (Nervous system disorders) | 6 | 1 | 1
Syncope (Nervous system disorders) | 4 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 3 | 0
Convulsion (Nervous system disorders) | 2 | 1 | 0
Loss of consciousness (Nervous system disorders) | 3 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 2 | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 2 | 0 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 1 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 1
Brain stem syndrome (Nervous system disorders) | 1 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 1
Cerebral artery occlusion (Nervous system disorders) | 0 | 0 | 1
Diabetic mononeuropathy (Nervous system disorders) | 0 | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 1 | 0 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0
Embolic stroke (Nervous system disorders) | 1 | 0 | 0
Facial palsy (Nervous system disorders) | 0 | 1 | 0
Grand mal convulsion (Nervous system disorders) | 1 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 1 | 0
Hydrocephalus (Nervous system disorders) | 0 | 1 | 0
Lacunar infarction (Nervous system disorders) | 0 | 1 | 0
Normal pressure hydrocephalus (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0
Radial nerve palsy (Nervous system disorders) | 1 | 0 | 0
Reversible ischaemic neurological deficit (Nervous system disorders) | 0 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | 0
Vascular headache (Nervous system disorders) | 1 | 0 | 0
Abortion spontaneous incomplete (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Major depression (Psychiatric disorders) | 0 | 2 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Anxiety disorder (Psychiatric disorders) | 0 | 0 | 1
Hypnagogic hallucination (Psychiatric disorders) | 0 | 0 | 1
Mental disorder (Psychiatric disorders) | 0 | 1 | 0
Panic attack (Psychiatric disorders) | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 2 | 7 | 1
Nephrolithiasis (Renal and urinary disorders) | 2 | 5 | 1
Calculus ureteric (Renal and urinary disorders) | 3 | 1 | 1
Renal colic (Renal and urinary disorders) | 2 | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 1
Calculus urethral (Renal and urinary disorders) | 0 | 1 | 0
Diabetic nephropathy (Renal and urinary disorders) | 0 | 1 | 0
Postrenal failure (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 0 | 1 | 0
Stress urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 3 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 3 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 2 | 0
Colpocele (Reproductive system and breast disorders) | 1 | 1 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 1 | 0
Genital prolapse (Reproductive system and breast disorders) | 2 | 0 | 0
Breast calcifications (Reproductive system and breast disorders) | 1 | 0 | 0
Epididymal cyst (Reproductive system and breast disorders) | 0 | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 1
Fallopian tube cyst (Reproductive system and breast disorders) | 0 | 1 | 0
Menometrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 1 | 0 | 0
Uterine prolapse (Reproductive system and breast disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Vocal cord polyp (Reproductive system and breast disorders) | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Knee arthroplasty (Surgical and medical procedures) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 1 | 1
Hypertension (Vascular disorders) | 2 | 0 | 0
Arteriosclerosis (Vascular disorders) | 0 | 1 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0
Pelvic venous thrombosis (Vascular disorders) | 0 | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alogliptin 12.5 mg (N=1394) | Alogliptin 25 mg (N=1399) | Rescued: Alogliptin 25 mg (N=527)
Hypertension (Vascular disorders) | 207 | 203 | 85
Urinary tract infection (Infections and infestations) | 155 | 163 | 71
Upper respiratory tract infection (Infections and infestations) | 162 | 153 | 49
Nasopharyngitis (Infections and infestations) | 133 | 162 | 44
Influenza (Infections and infestations) | 113 | 132 | 42
Diarrhoea (Gastrointestinal disorders) | 108 | 115 | 53
Arthralgia (Musculoskeletal and connective tissue disorders) | 118 | 108 | 37
Back pain (Musculoskeletal and connective tissue disorders) | 102 | 111 | 46
Headache (Nervous system disorders) | 90 | 105 | 40
Bronchitis (Infections and infestations) | 94 | 111 | 26
Dyslipidaemia (Metabolism and nutrition disorders) | 80 | 80 | 30
Oedema peripheral (General disorders) | 70 | 84 | 30
Cough (Respiratory, thoracic and mediastinal disorders) | 84 | 72 | 27
Pain in extremity (Musculoskeletal and connective tissue disorders) | 67 | 80 | 32
Pharyngitis (Infections and infestations) | 67 | 69 | 27
Sinusitis (Infections and infestations) | 70 | 64 | 23
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 54 | 62 | 28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.